CLINICAL TRIAL: NCT07045792
Title: Investigating the Effects of Body Awareness Therapy on Functional Capacity, Balance, Sleep Quality and Psychological State in Young Adults With High Stress Levels: A Randomized Controlled Trial
Brief Title: Body Awareness Therapy in High Stressed Young Adults: Effects on Function, Balance, Sleep and Mood
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Yasemin KARAASLAN, Principal Researcher, Head of Physiotherapy and Rehabilitation Department, Hatay Mustafa Kemal University, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BFT2025-01
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Stress; Psychological Factors; Sleep; Postural Balance
Keywords: Body Awareness Therapy; Stress Levels; Psychological Stress; Balance; Sleep Quality; Functional Capacity; Physical Therapy; Postural Balance
MeSH Terms: conditions — Stress, Psychological; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No intervention
- Intervention Group (Experimental): Body Awareness Therapy
  Interventions: Procedure: Body Awareness Therapy

INTERVENTIONS:
Procedure: Body Awareness Therapy — Individuals trained for body awareness therapy.
  Arms: Intervention Group

SUMMARY:
Body Awareness Therapy (BAT) is a holistic approach to human movement that considers the physical, physiological, psychological, and existential aspects of human existence. This planned randomized controlled study will be conducted on young adults with high stress levels. One group will be subjected to BAT and the other group will be the control group. The BAT exercises will be performed in supine, sitting and standing positions. In the BAT group, the exercises will be performed as a group exercise, not individually. After the initial evaluations in both the BAT and control groups, a re-evaluation will be performed at the end of 8 weeks. Functional capacity will be assessed with the 6-minute walk test, static balance with the single-leg balance test (eyes open-eyes closed), dynamic balance with the Y-balance test, psychological status with the Depression-Anxiety-Stress Scale-21 (DASS-21), and sleep quality with the Pittsburgh Sleep Quality Scale. BAT will be performed 2 days per week for 8 weeks and will be continued progressively. This study will examine the effects of BaT on functional capacity, balance, sleep quality, and psychological state in young adults with high stress levels.

DETAILED DESCRIPTION:
This study will follow a randomized controlled trial design. The study will be conducted in young adults at the Faculty of Health Sciences, Hatay Mustafa Kemal University.

The estimation of the sample size was conducted by calculating the requirement of a sample of 52 participants (26 per group) to achieve 80% power with an effect size of d = 0.80, α = 0.05, type I error, and β = 0.20, type II error. To account for potential exclusions from the study and data loss during the implementation process, the reserve participant rate was calculated to be 20%. Therefore, following the analysis, it was determined that the study would be conducted with a total of 62 participants, with 31 participants allocated to each group.

All assessments will be conducted in person by the research team. A comprehensive evaluation of the descriptive information, functional capacity, balance, sleep quality, and psychological status of the study participants is warranted.

Treatment Program Individuals in the BAT group will train 2 days per week for 8 weeks. The training will be conducted by a person who has received BAT training at levels A, B, C and D at the Swedish Institute of Body Awareness (Institutet Basal Kroppskännedom).

Those in the control group will not receive any training and will remain on the waiting list. These patients will also be assessed at baseline and after 8 weeks. In this group, BAT will be applied to the students who want to receive the training after the last measurements.

Body Awareness Therapy Exercises consist of awareness exercises in the supine, sitting, standing, and walking positions: Considering eight weeks, the training is designed to progress gradually after every two weeks. The BAT exercises are done in groups of 6 people.

The BAT program consists of 40 minutes of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Be between 20 and 30 years old
* Be literate
* Score 10 or above on the stress subscale of the Depression Anxiety Stress Scale -21
* Be willing to participate in the study voluntarily

Exclusion Criteria:

* Individuals with orthopedic, neurological, rheumatological, psychiatric, mental, or any systemic chronic diseases
* Those with cardiac problems that may prevent exercise
* Those suspected of being pregnant
* Individuals with malignancy
* Individuals with active infection
* Those who do not regularly attend the treatment program

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
6-Minute Walk Test | 8 weeks
  They will be asked to walk as fast as they can down a 30-meter straight corridor for 6 minutes.
Single Leg Stance Test | 8 weeks
  The maximum time that individuals can stand on one leg with eyes open and closed will be recorded.
Y Balance Test | 8 weeks
  During the test, 3 trials will be performed for each leg and the best score will be recorded (right anterior, left anterior, right posteromedial, left posteromedial, right posterolateral, left posterolateral). The maximum reach distance was recorded for each consecutive trial.
Depression Anxiety Stress Scale - 21 | 8 weeks
  Psychological status will be evaluated. The total score for each heading ranges from 0 to 21. Higher total scores indicate higher depression, higher anxiety, and higher stress levels.
Pittsburgh Sleep Quality Index | 8 weeks
  Sleep quality will be evaluated. The 19 items measure seven subcomponents. Each question is scored between "0" and "3". The total score (0-21) is obtained by adding the seven subscores. According to the total score, those with a score of 5 and below are interpreted as having good sleep quality, and those with a score above 5 are interpreted as having poor sleep quality.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire - Short Form | 8 weeks
  Physical activity will be evaluated. Individuals with less than 600 METs of physical activity per week are classified as "inactive", individuals with 600 to 3000 METs per week are classified as "minimally active", and individuals with more than 3000 METs per week are classified as "very active".

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal University, Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Hatay, Antakya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
At the end of the study, with the acceptance of the article, the data requested by the reader can be shared with the approval of the authors.